CLINICAL TRIAL: NCT02938754
Title: Motor and Cognitive Training With the Rehabilitation Gaming System for Patients Affected by Cerebral Palsy
Brief Title: Rehabilitation Gaming System for Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Pompeu Fabra (Other)
Responsible Party: Principal Investigator, Paul Verschure, PhD, Universitat Pompeu Fabra
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VR for Cerebral Palsy
Record Dates: First submitted 2016-06-22; First posted 2016-10-19 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Cerebral Palsy; Movement Disorder
Keywords: Hemiparesis; Functional independence; Virtual Rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Movement Disorders; Paresis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VR-based motor training (Experimental): Subjects will perform 3 different training protocols in Virtual Reality that imply performing tasks of vertical and planar reaching and hitting spheres, or hockey pucks, spaced at different time, speed and color.
  Interventions: Behavioral: VR-based motor training
- Conventional Therapy (Active Comparator): Subjects will perform conventional rehabilitation tasks for the upper-extremities that imply vertical and planar reaching movements.
  Interventions: Behavioral: Conventional Therapy

INTERVENTIONS:
Behavioral: VR-based motor training — Subjects will perform 3 different training protocols in Virtual Reality that imply performing tasks of vertical and planar reaching and hitting spheres, or hockey pucks, spaced at different time, speed and color.
  Arms: VR-based motor training
Behavioral: Conventional Therapy — Subjects will perform conventional rehabilitation tasks for the upper-extremities that imply vertical and planar reaching movements.
  Arms: Conventional Therapy

SUMMARY:
In this study the investigators evaluate the effectivity of Virtual Reality-based rehabilitation protocols for preventing motor deterioration in patients with cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Children and Adult patients between 12- 50 years old diagnosed with CP according to Gross Motor Function Classification System (GMFCS). Level of disability between I and IV.
* Ashworth modified clinical scale < 3 (Ashworth, 1964, Bohannon Bohannon and Smith, 1987).

Exclusion Criteria:

* Severe visual impairment.
* Severe cognitive impairment such as mental retardation which impedes the understanding of the task.

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in motor function of the affected extremity as measured by MACS clinical scale | Change from Baseline to week 5 (End of Treatment)

SECONDARY OUTCOMES:
Change in attention and visuo-perceptive and visuo-constructional apraxia as measured by the WAIS-III scale | Change from Baseline to week 5 (End of Treatment)
Change in motor function of the affected extremity as measured by the Box and Blocks clinical scale | Change from Baseline to week 5 (End of Treatment)
Change in the amount of use of the affected arm during training as measured by the Virtual Reality system | Change from Baseline to week 5 (End of Treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Paul FMJ Verschure, PhD, Principal Investigator — Center of Autonomous Systems and Neurorobotics
Locations (1):
- Universitat Pompeu Fabra, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cameirao MS, Badia SB, Duarte E, Frisoli A, Verschure PF. The combined impact of virtual reality neurorehabilitation and its interfaces on upper extremity functional recovery in patients with chronic stroke. Stroke. 2012 Oct;43(10):2720-8. doi: 10.1161/STROKEAHA.112.653196. Epub 2012 Aug 7. PMID 22871683
- [Background] Wittenberg GF. Neural plasticity and treatment across the lifespan for motor deficits in cerebral palsy. Dev Med Child Neurol. 2009 Oct;51 Suppl 4:130-3. doi: 10.1111/j.1469-8749.2009.03425.x. PMID 19740220